CLINICAL TRIAL: NCT06971016
Title: "Effectiveness of Mulligan Mobilization Technique and Proprioceptive Exercises Among Patients With Knee Osteoarthritis in Karachi" The Study Will Include Individuals Diagnosed With Knee OA, Aged 40 Years and Above, Clinically Diagnosed Mild to Moderate Primary OA in Knee. Participants Will be Recruited From a Physical Therapy Clinic, and Will be Screened for Inclusion and Exclusion Criteria. Inclusion Criteria Will Include Diagnosed Cases of Knee OA With Mild to Moderate Grade of OA (According to Kellgren and Lawrence Scale) and the Ability to Walk Without Assistive Device for at Least 50 Feet
Brief Title: "Effectiveness of Mulligan Mobilization Technique and Proprioceptive Exercises Among Patients With Knee Osteoarthritis"
Acronym: MWMPETKOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Center (Other)
Responsible Party: Principal Investigator, Muhammad Atif Khan, Principal Investigator, National Healthcare Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUC/MKT/IND/SP/03/327; Lincoln University College (Other: Lincoln University College)
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis; Mulligan Mobilization; Proprioceptive training; Pain; Functional Status; Knee Managment
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Total 60 subjects will be selected by simple random sampling and equally divided into 3 groups:
  Experimental Group A=Proprioceptive exercises group Experimental Group B=Mulligan Mobilization Technique Group Control Group C= Traditional Physical Therapy. The study will follow a pre-test and post-test design, with assessments to be conducted at baseline, immediately after intervention and 10-weeks follow-up.
  Study will be continued for 10 weeks and a total number of 30 treatment sessions will be given to each patient with 3 sessions per week.
  Assessment of the patients will be done at the beginning of 1st Session day and at the end of treatment of 30th Session day.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Exercises (Experimental): Proprioceptive exercises aim to enhance an individual's ability to perceive body position and movement in space, improving balance, stability, and injury prevention. These exercises have shown significant benefits for various populations, including institutionalized older adults, where they improved functional mobility, balance, gait, and reduced fall risk.
  Interventions: Other: Proprioceptive Exercises
- Mulligan Mobilization Technique (Active Comparator): The Mulligan Mobilization Technique, specifically Mobilization with Movement (MWM), is an effective manual therapy approach for treating musculoskeletal conditions. In knee osteoarthritis treatment, Mulligan mobilization was found to be more effective than Maitland technique in alleviating pain and improving function scores. The technique can be combined with other therapeutic measures such as conventional treatments and exercises for optimal results. Overall, Mulligan Mobilization Technique emerges as a promising intervention for various musculoskeletal conditions, offering pain relief and functional improvement.
  Interventions: Other: Mulligan Mobilization technique
- Placebo (Placebo Comparator): Traditional Physical Therapy
  Interventions: Other: Traditional Physical therapy

INTERVENTIONS:
Other: Mulligan Mobilization technique — i. Mulligan Mobilization for Medial Glide: During the treatment, the patient will be positioned in a prone (face-down) posture. To execute a medial glide, the therapist will position themselves on the side opposite to the target knee. They will place a belt around the patient's waist and lower leg, aligning the upper edge of the belt with the margin of the tibial joint. Using one hand to stabilize the thigh above the knee and the other hand to support the lower leg, the therapist will apply a medial force to the knee using the belt. The therapist will then instruct the patient to flex their knee while maintaining the glide.
  ii. Mulligan Mobilization for Lateral Glide: To administer a lateral glide to the knee, the therapist will position themselves next to the affected knee. They will employ the belt to facilitate the glide by applying force from the opposite side.
  Arms: Mulligan Mobilization Technique
Other: Proprioceptive Exercises — i. One leg balance- It requires flexing the opposite leg at the knee, hip, and ankle while standing on the affected foot. This position will be hold for one minute (60 seconds), followed by rest for 10 to 20 seconds, then continue this process twice more. Three repetitions of the same exercise will be performed with the unaffected leg after a brief break.
  ii. Blind advanced one leg balance- The task will resemble one-legged balance, but the participant will be required to close their eyes while executing the routine, and then repeat it two more times.
  iii. Toe walking- In this activity, the participant will be instructed to walk a 20-meter distance while balancing on their toes with their toes pointing straight ahead. They will then be asked to walk the same distance again, but this time with their toes pointing outward. After a brief rest, the entire procedure will be repeated once more.
  Arms: Proprioceptive Exercises
Other: Traditional Physical therapy — • Stretching of the Gastrocnemius and Soleus Muscles
  * Frequency: 3-5 times per week.
  * Intensity: Stretch to the point of mild discomfort, not pain.
  * Time: Hold each stretch for 30 seconds and repeat 3 times on each leg.
  * Type: Static stretching. Gastrocnemius Stretch: Stand facing a wall with one foot forward (slightly bent) and the other foot back (straight). Press the back heel into the floor and lean forward to feel the stretch in the calf.
  Soleus Stretch: From the same position, slightly bend the back knee while keeping the heel on the ground to target the lower calf (soleus muscle).
  • Stretching of the Hamstrings
  * Frequency: 3-5 times per week.
  * Intensity: Stretch to a tolerable point of tension without causing pain.
  * Time: Hold each stretch for 30 seconds and repeat 3 times on each leg.
  * Type: Static stretching. Seated Hamstring Stretch: Sit on the floor with one leg straight and the other bent.
  Arms: Placebo

SUMMARY:
This research analyzes the effectiveness of Mulligan mobilization in comparison to proprioceptive exercises for treating patients with mild to moderate Knee osteoarthritis whose condition falls under Kellgren and Lawrence grading system Grades 2 and 3. The current study evaluates these therapeutic approaches as a combined method during a 10-week assessment period which incorporates pain intensity measures, movement analysis and functional activities and balance performance together with quality of life improvement. The study implements a preliminary test followed by standardized evaluation tests to establish robust data for Knee osteoarthritis physical therapy strategies.

The study population will include individuals diagnosed with knee OA, aged 40 years and above, clinically diagnosed mild to moderate primary OA in knee. Participants will be recruited from a physical therapy clinic, and will be screened for inclusion and exclusion criteria. Inclusion criteria will include diagnosed cases of knee OA with mild to moderate Grade of OA (According to Kellgren and Lawrence Scale) and the ability to walk without assistive devices for at least 50 feet.

A total of 60 subjects will be chosen equally for three groups (Experimental Group A=Proprioceptive Exercises group), (Experimental Group B=Mulligan Mobilization Technique Group), and (Control Group C= Traditional physical therapy). Double blinding randomized selection through simple random sampling will determine all participants. Study will continue for 10 weeks and a total number of 30 treatment sessions will be given to each patient with 3 sessions per week. Session lasting an average of 40 minutes to an hour each. Assessment of the patients will be done at the beginning of 1st Session day and at the end of treatment of 30th Session day. The research site for this investigation is Physiotherapy Out-Patient Department at National Healthcare Centre, Karachi-Pakistan.

DETAILED DESCRIPTION:
The research examines the effectiveness comparison between Mulligan Mobilization Technique and Proprioceptive Exercises for knee OA patients by adopting the following illustrated conceptual framework.

The study's independent variable consists of both Mulligan Mobilization Technique and Proprioceptive Exercises as treatment interventions. The evaluation tools include Numeric Pain Rating Scale (NPRS), Universal Goniometer, Knee Injury and OA Outcome Score (KOOS), Berg Balance Scale (BBS) and Quality of Life Short Form (SF-36) for assessing pain, range of motion, functional status, balance and quality of life respectively.

The research's experiment expects the independent treatment to modify the analyzed outcomes. The pre-test and post-test experimental setup will assess how well the intervention treatments affect the dependent variables. Two treatments known as Mulligan Mobilization Technique with Proprioceptive Exercises will be assessed for their effectiveness in treating knee OA patients throughout the study. The study will evaluate the effect of age together with gender and body mass index (BMI) as well as disease severity on outcomes from different interventions.

CONSENT FORM (ENGLISH) Title of Study: Effectiveness of Mulligan Mobilization Technique and Proprioceptive Exercises among Patients with Knee Osteoarthritis in Karachi

Introduction: You are being invited to participate in a research study. Please read this form carefully and feel free to ask any questions you may have before agreeing to participate.

Purpose of the Study: The purpose of this study is to compare the effectiveness of Mulligan Mobilization Technique versus Proprioceptive Exercises on pain, range of motion, functional status, balance and quality of life among patients with knee OA.

Procedures: If you agree to participate in this study, you will be asked to complete a series of questionnaires to evaluate your pain, range of motion, functional status, balance and quality of life. You will also receive either Mulligan Mobilization Technique, Proprioceptive Exercises or Traditional Physical Therapy depending on the group you are randomly assigned to Mulligan Mobilization Technique is a manual therapy technique that aims to improve joint mobility and reduce pain. Proprioceptive Exercises are exercises that focus on improving balance and joint position sense. The treatment will be performed by a licensed physical therapist who has been trained to perform both techniques. You will receive 30 sessions of treatment over a period of ten weeks. Each session will last approximately 45 minutes.

Risks and Benefits: There are no anticipated risks associated with participating in this study. However, some participants may experience temporary pain or discomfort during the treatment sessions. The benefits of participating in this study include the potential to improve pain, range of motion, functional status, balance and quality of life among patients with knee OA. Participants are requested not to perform other treatment or take any painkillers during the period of intervention and evaluation.

Confidentiality: Your participation in this study will be kept confidential. Your personal information will be kept in a secure location and will only be accessible to the researchers involved in the study.

Voluntary Participation: Your participation in this study is completely voluntary. You have the right to withdraw from the study at any time without any penalty.

Contact Information: If you have any questions or concerns about the study, please feel free to contact Muhammad Atif Khan (Principal Investigator) at 0092-332-2281028 or mak_physio@yahoo.com.

Consent: By signing below, you acknowledge that you have read and understood the information provided in this form, and you voluntarily agree to participate in the study.

Participant Signature: ____________________________ Date: _________________

Researcher Signature: _____________________________ Date: _________________

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include diagnosed cases of knee OA with mild to moderate Grade of OA (According to Kellgren and Lawrence Scale)
* Ability to walk without assistive devices for at least 50 feet.

Exclusion Criteria:

* Patients have Kellgren and Lawrence <grade 2 or above grade 3
* History of knee surgery, knee joint replacement
* Patients have been administered corticosteroid injections in last six months - - - History of mental illness, autoimmune disorder, neurological or orthopedic conditions affecting the lower limbs
* Presence of any other conditions that may affect balance or gait.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 10 weeks
  The KOOS exists to measure both brief and persistent symptoms together with actual functions of people who have knee ligament damage or osteoarthritis. General healthcare providers rely on the KOOS tool as well as research investigators to track patient health evolution through registries and clinical use. This evaluation instrument contains five distinct subcategories which assess Pain as well as Symptoms alongside Activities of Daily Living (ADL) and Sports and Recreation Function (Sport/Rec) and Knee-Related Quality of Life (QOL). Each subscale in KOOS receives scoring on a 5-point Likert scale before the scores transform into a 0 to 100 scale representing extreme symptoms to no symptoms.
Universal Goniometer | 10 weeks
  Physical therapy practitioners use universal goniometers (UG) to conduct goniometry which stands as an necessary technique for measuring joint range of motion (ROM). A two-armed handheld device provides stable measured results through valid procedures if users adhere to specific placement protocols.
Numeric Pain Rating Scale (NPRS) | 10 weeks
  Through NPRS participants rate their pain levels on a 0 to 10 scale by choosing numbers that show no pain at 0 and maximum pain at 10. The pain intensity score is determined by the number that the participant selects.
Berg Balance Scale (BBS) | 10 weeks
  The Berg Balance Scale stands as a common instrument which evaluates testing both static and dynamic balance levels. The BBS created by Katherine Berg during 1989 contains 14 specific tasks that measure both sitting and standing and dynamic balance abilities of patients. Therapy participants receive scores ranging from 0 to 4 on each task distributed across a total rate of 56 points in the assessment process.

SECONDARY OUTCOMES:
Quality of Life Short Form (SF-36) | 10 weeks
  The SF-36 provides a full instrument for measuring health-related quality of life through 36 items with eight domain categories including Physical Function (PF) and Role Physical (RP) and Bodily Pain together with General Health (GH) as well as Vitality (VT) and Social Function (SF) and Role Emotional (RE) and Mental Health (MH). The SF-36 organizes its measures under two main domains named Physical Component Summary and Mental Component Summary which serve as scoring categories. Standard deviation scores follow norms that use 50 as mean and 10 as standard deviation to achieve population-wide evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Atif Khan, PhD Scholar, Principal Investigator — National Healthcare Center
Locations (1):
- National Healthcare Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations and the need to protect participant confidentiality, individual participant data will not be shared. The informed consent obtained from participants does not include permission for data sharing with external researchers.

REFERENCES:
- [Background] Rao RV, Balthillaya G, Prabhu A, Kamath A. Immediate effects of Maitland mobilization versus Mulligan Mobilization with Movement in Osteoarthritis knee- A Randomized Crossover trial. J Bodyw Mov Ther. 2018 Jul;22(3):572-579. doi: 10.1016/j.jbmt.2017.09.017. Epub 2017 Sep 28. PMID 30100279
- See also: this the evidence which help to formulate the study protocol — https://pubmed.ncbi.nlm.nih.gov/30100279/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT06971016/Prot_SAP_ICF_000.pdf